CLINICAL TRIAL: NCT01681927
Title: Study of Idiopathic Edema
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, John Maesaka, MD, Acting Chief of Nephrology and Hypertension, Winthrop University Hospital
Other Study IDs: 220488-4; WUH 350-595 (Other: Winthrop-University Hospital)
Record Dates: First submitted 2012-08-08; First posted 2012-09-10 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Idiopathic Edema Nocturia
Keywords: idiopathic edema nocturia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1.4kg wt gain 8AM -10 PM: Complete a questionnaire. Measure and record weight in AM and PM.Record for one week,number of times urinated after bedtime and before waking up.
- >1.4kg wt gain 8AM - 10PM no nocturia.: Complete a questionnaire. Measure and record weight in AM and PM.Record for one week,number of times urinated after bedtime and before waking up.
- > 1.4 kg wt gain 8AM -10PM with nocturia: Complete a questionnaire. Measure and record weight in AM and PM. Record the number of times and collect all urine passed overnight in separate containers for one week.Collection of blood and interstitial fluid samples, fluorescein dye angiography, and bioimpedance study.

SUMMARY:
Idiopathic edema (IE) is an ill-defined syndrome of uncertain etiology that occurs virtually exclusively in women. It has also been referred to as cyclical edema, periodic edema, fluid retention syndrome and orthostatic edema.

The present studies were designed to 1. Improve our ability to identify patients with idiopathic edema by extending the clinical criteria from an increase in weight of > 1.4 kg between 8 AM to 10 PM to the inclusion of nocturia, a very important component to the history. Additional aims are to: 2. Demonstrate orthostatic weight gain with or without edema in idiopathic edema and autonomic failure that will identify a greater number of patients suffering from variable degrees of weight gain and compare to controls or other conditions associated with edema. The study will focus mainly on subjects with polycystic ovaries and autonomic failure. 3. Provide a reasonable course of therapy that is presently not well defined. 4. Provide evidence that orthostatic edema or weight gain has two common etiologies, a. an increase in vascular membrane as in idiopathic edema and b. pooling of blood in the lower extremities in autonomic failure due to a lack of vascular tone.

DETAILED DESCRIPTION:
All postmenarchal female patients over the age of 14 years will be eligible to enter the study except for the following exclusions: serum creatinine > 2.0 mg/dl, patients with diabetes insipidus-nephrogenic and central, those on lithium therapy and diuretics that cannot be held for 3 days. Subjects under the age of 18 will be asked tp complete the questionnaire, which requires that the subject record the weights at 8 AM and 10 PM and whether they get up at night to urines. If they gain more than three pounds during the day and get up at night to urinate, they will be asked to keep a record of their weights and the number of times they get up at night to urinate for one week. A consent form for patients below the age of 18 has been developed for this age-group. Patients will be recruited from referrals from the different subspecialty groups in the Winthrop Hospital system, mainly pediatric endocrinology, obstetric and gynecology, neurology, ophthalmology, cardiology and gastroenterology practices.

The subjects will be placed in the following groups:

Group I: nonedematous patients

1. polycystic ovaries
2. autonomic failure-male and female
3. Age and gender matched normals Group II-Edema not meeting criteria for idiopathic edema

1.Congestive heart failure 2.Cirrhosis of liver 3.Nephrosis 4.Pregnancy 5.Pre eclampsia 6.Unknown cause of edema, such as obesity. Group III-Orthostatic weight gain of > 3 lbs between 8 AM and 10 PM with nocturia

1. Idiopathic edema, include patients in Group I-fluctuations in weight/nocturia
2. Autonomic failure, include patients in Group I-fluctuations in weight/nocturia

Group III subjects will undergo the following procedures:

1. Record weights in pajamas before bedtime and after excreting first urine upon arising in the morning for 1 week.
2. Record the number of times they get up to urinate and collect all urines passed overnight in separate containers, including urine excreted upon arising in the morning. The patient will record the time and date on each container provided for this purpose.

24 hour study:

1. Blood will be collected after waking up the following morning and at 7 PM the same day. Blood will be analyzed for renal profile, renin, aldosterone, uric acid, phosphorus
2. All urines excreted from the time after arising in the morning and collected in separate containers throughout the following 24 hours and the times of collection noted. The urines will be analyzed for osmolality, sodium, potassium, creatinine, uric acid, urea and phosphorus.

Bioimpedance Studies:

Patients in group III will have bioimpedance studies performed in the morning upon arising and in the evening to determine any change in body composition, i.e. change in volume of extracellular, intracellular and total body water.

Collection of Interstitial Fluid:

In selected patients, an 18g needle will be placed subcutaneously in the mid-thigh and the interstitial fluid collected by gravity to obtain 2-3 ml of fluid for analysis in late afternoon. A blood sample will be obtained after completion of the sampling of edema fluid. The serum will be analyzed for renal profile, total protein, albumin and electrophoresis. The interstitial fluid will analyzed for renal profile, osmolality, total protein, albumin and electrophoresis.

Fluorescein dye studies:

Patients in Group III and selected patients with polycystic ovaries without edema over the age of 18 years will undergo a standard ophthalmologic fluorescein dye test to detect any increase in vascular endothelial permeability. Patients with diabetes mellitus will be excluded from this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects gaining > 1.4 kg and nocturia

Exclusion Criteria:

* those not gaining > 1.4 kg and without nocturia

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with idiopathic edema
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Orthostatic weight exceeding 1.4 kg/day | 1 day
  the subject will record weights upon arising and before retiring at night.

SECONDARY OUTCOMES:
Nocturia | overnight
  The subject will record and save all urines excreted after retiring for the night and upon arising in the morning.

CONTACTS AND LOCATIONS:
Overall Officials: John K Maesaka, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop-University Hospital, Mineola, New York, United States